CLINICAL TRIAL: NCT02029495
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Study to Evaluate the Efficacy, Safety and Effect on Radiographic Progression of Brodalumab in Subjects With Psoriatic Arthritis: AMVISION-1
Brief Title: Study of Efficacy, Safety and Effect on Radiographic Progression of Brodalumab in Subjects With Psoriatic Arthritis
Acronym: AMVISION-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20090406; 2013-003554-25 (EudraCT Number)
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; Brodalumab; AMG 827
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — brodalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 210 mg brodalumab (Experimental): Administered via subcutaneous injections
  Interventions: Drug: 210 mg brodalumab
- 140 mg brodalumab (Experimental): Administered via subcutaneous injection
  Interventions: Drug: 140 mg brodalumab
- Placebo (Placebo Comparator): Administered via subcutaneous injection until week 24.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 210 mg brodalumab — 210 mg brodalumab administered via subcutaneous injection
  Other Names: AMG 827
  Arms: 210 mg brodalumab
Drug: 140 mg brodalumab — 140 mg brodalumab administered via subcutaneous injection
  Other Names: AMG 827
  Arms: 140 mg brodalumab
Drug: Placebo — Placebo administered via subcutaneous injection until week 24.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of brodalumab, compared to placebo, in subjects with psoriatic arthritis.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of brodalumab, compared to placebo, in subjects with psoriatic arthritis. The key secondary objective is to evaluate the efficacy of brodalumab compared to placebo at week 16 and week 24. The safety objective of this study is to evaluate the safety profile of brodalumab in subjects with psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of psoriatic arthritis (by the Classification of Psoriatic Arthritis criteria (CASPAR), with ≥ 3 tender and ≥ 3 swollen joints (excluding the distal interphalangeal joints)).
* Subjects must have at least 1 psoriatic skin lesion as well as either ≥ 1 erosion on a centrally read radiograph or an elevated CRP.

Exclusion Criteria:

* Subject has known history of active tuberculosis.
* Subject has a planned surgical intervention between baseline and the week 52 evaluation.
* Subject has an active infection or history of infections.
* Subject has any systemic disease (eg, renal failure, heart failure, hypertension, liver disease, diabetes, anemia) considered by the Investigator to be clinically significant and uncontrolled.
* Subject has any concurrent medical condition or electrocardiogram (ECG) abnormality that, in the opinion of the investigator, could cause this study to be detrimental to the subject.
* Subject has severe depression measured by Personal Health Questionnaire Depression Scale (PHQ-8) or suicidal ideation/behavior as measured by and Columbia Suicide Severity Rating Scale (e-CSSRS)
* Subject has a history or evidence of psychiatric disorder or substance abuse considered by the Investigator to pose a risk to subject safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (131):
- United States (43):
  - Research Site, Huntsville, Alabama
  - Research Site, Tuscaloosa, Alabama
  - Research Site, Peoria, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Mather, California
  - Research Site, Murrieta, California
  - Research Site, Palm Desert, California
  - Research Site, Tustin, California
  - Research Site, Upland, California
  - Research Site, Jupiter, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Tampa, Florida
  - Research Site, Gainesville, Georgia
  - Research Site, Meridian, Idaho
  - Research Site, Springfield, Illinois
  - Research Site, Bowling Green, Kentucky
  - Research Site, Somerset, Kentucky
  - Research Site, Frederick, Maryland
  - Research Site, Wheaton, Maryland
  - Research Site, Worcester, Massachusetts
  - Research Site, Lansing, Michigan
  - Research Site, Eagan, Minnesota
  - Research Site, Omaha, Nebraska
  - Research Site, Clifton, New Jersey
  - Research Site, Great Neck, New York
  - Research Site, Lake Success, New York
  - Research Site, New York, New York
  - Research Site, Plainview, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Bend, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Hixson, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Danville, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Beckley, West Virginia
  - Research Site, Bridgeport, West Virginia
  - Research Site, Glendale, Wisconsin
- Belgium (2):
  - Research Site, Hasselt
  - Research Site, Leuven
- Bulgaria (3):
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
- Canada (5):
  - Research Site, Calgary, Alberta
  - Research Site, Toronto, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Trois-Rivières, Quebec
- Czechia (6):
  - Research Site, Brno
  - Research Site, České Budějovice
  - Research Site, Ostrava-Trebovice
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Uherské Hradiště
- Estonia (2):
  - Research Site, Pärnu
  - Research Site, Tallinn
- France (6):
  - Research Site, Cahors
  - Research Site, Orléans
  - Research Site, Rennes
  - Research Site, Saint-Etienne
  - Research Site, Toulouse
  - Research Site, Tours
- Greece (3):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Thessaloniki
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Esztergom
  - Research Site, Nyíregyháza
  - Research Site, Székesfehérvár
  - Research Site, Szolnok
- Italy (7):
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Pavia
  - Research Site, Roma
  - Research Site, Roma (RM)
  - Research Site, Rome
  - Research Site, Verona
- Mexico (7):
  - Research Site, Mexicali, Baja California Norte
  - Research Site, Chihuahua City, Chihuahua
  - Research Site, León, Guanajuato
  - Research Site, Guadalajara, Jalisco
  - Research Site, Distrito Federal, Mexico
  - Research Site, Ciudad Obregón, Sonora
  - Research Site, Mérida, Yucatán
- Poland (10):
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Katowice
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Stalowa Wola
  - Research Site, Świdnik
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Russia (7):
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- Slovakia (4):
  - Research Site, Banská Bystrica
  - Research Site, Lučenec
  - Research Site, Rimavská Sobota
  - Research Site, Žilina
- Spain (10):
  - Research Site, Córdoba, Andalusia
  - Research Site, Granada, Andalusia
  - Research Site, Seville, Andalusia
  - Research Site, Barcelona, Catalonia
  - Research Site, L'Hospitalet de Llobregat, Catalonia
  - Research Site, Sabadell, Catalonia
  - Research Site, Mérida, Extremadura
  - Research Site, A Coruña, Galicia
  - Research Site, Madrid, Madrid
  - Research Site, Villajoyosa, Valencia
- Switzerland (4):
  - Research Site, Basel
  - Research Site, Geneva
  - Research Site, Lausanne
  - Research Site, Zurich
- United Kingdom (6):
  - Research Site, Birmingham
  - Research Site, Glasgow
  - Research Site, Hull
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 210 mg Brodalumab | 140 mg Brodalumab | Placebo
Started | 159 | 158 | 161
Completed | 158 | 158 | 159
Not Completed | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 210 mg Brodalumab | 140 mg Brodalumab | Placebo | Total
Number analyzed (Participants) | 159 | 158 | 161 | 478
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 144 | 138 | 145 | 427
  >=65 years | 15 | 20 | 16 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (12.24) | 49.9 (12.80) | 48.1 (11.79) | 49 (12.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 80 | 80 | 230
  Male | 89 | 78 | 81 | 248
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 0 | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 155 | 152 | 152 | 459
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 6 | 5 | 13
Region of Enrollment [Number; unit: participants]
  Russian Federation | 22 | 22 | 27 | 71
  Hungary | 5 | 6 | 4 | 15
  United States | 35 | 37 | 35 | 107
  United Kingdom | 6 | 3 | 6 | 15
  Switzerland | 1 | 6 | 5 | 12
  Spain | 10 | 4 | 7 | 21
  Greece | 2 | 2 | 2 | 6
  Canada | 4 | 3 | 2 | 9
  Czech Republic | 2 | 8 | 9 | 19
  Belgium | 0 | 0 | 2 | 2
  Poland | 50 | 45 | 44 | 139
  Italy | 2 | 5 | 2 | 9
  Mexico | 5 | 3 | 4 | 12
  Slovakia | 5 | 5 | 5 | 15
  France | 4 | 2 | 2 | 8
  Bulgaria | 2 | 4 | 3 | 9
  Estonia | 4 | 3 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: American College of Rheumatology (ACR) 20 Response
Description: An ACR20 response is defined as at least 20% improvement of tender and swollen joint counts combined with at least 20% improvement in at least 3 of the following 5 parameters: Patients Global Assessment, PtGA of disease activity, patient's assessment of pain, Health Assessment Questionnaire-Disability Index (HAQ-DI), and either Erythrocycte sedimentation rate (ESR) or C-Reactive protein (CRP) (ACR components).
Time Frame: 16 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 210 mg Brodalumab | 140 mg Brodalumab | Placebo
Number analyzed (Participants) | 121 | 118 | 122
percentage of participants | 0 [0 to 0] | 21.8 [10.6 to 33.1] | 36.5 [22.8 to 45.3]

2. Secondary Outcome: Psoriasis Area and Severity Index (PASI)75
Description: PASI75 indicates that the subject has had a response of a 75% reduction on the severity of the psoriasis area based of off effected area size, erythema, scaling, and itching.
Time Frame: 16 Weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 210 mg Brodalumab | 140 mg Brodalumab | Placebo
Number analyzed (Participants) | 61 | 72 | 60
percentage of participants | 70.3 [57.6 to 82.9] | 55.6 [27.9 to 56.6] | 0 [0 to 0]

ADVERSE EVENTS:
Arm/Group | 210 mg Brodalumab | 140 mg Brodalumab | Placebo
Serious Adverse Events (participants affected / at risk) | 10/158 | 5/158 | 4/159
Other Adverse Events (participants affected / at risk) | 84/158 | 79/158 | 71/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 210 mg Brodalumab (N=158) | 140 mg Brodalumab (N=158) | Placebo (N=159)
Urosepsis (Infections and infestations) | 1 | 0 | 0
Squimos Cell Carcinoma of the Vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Major Depression (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Dizziness (General disorders) | 0 | 1 | 0
Lens Dislocation (Eye disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Drug reaction with Eosinaphilia and Systematic symptoms (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral Disc protusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Eye Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Iris Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Keratorhexis (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 210 mg Brodalumab (N=158) | 140 mg Brodalumab (N=158) | Placebo (N=159)
Nasopharyngitis (Infections and infestations) | 24 | 28 | 7
Upper Respiratory tract Infection (Infections and infestations) | 9 | 9 | 8
Diarrheoa (Gastrointestinal disorders) | 2 | 5 | 3
Headache (Nervous system disorders) | 5 | 4 | 3
Hypertension (Vascular disorders) | 10 | 2 | 3
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 3 | 5
bronchitis (Infections and infestations) | 6 | 5 | 2
Sinusitis (Infections and infestations) | 3 | 3 | 2
Rhinitis (Infections and infestations) | 4 | 0 | 3
urinary Tract Infection (Infections and infestations) | 2 | 0 | 3
Viral infection (Infections and infestations) | 2 | 0 | 0
gastroenteritis (Infections and infestations) | 1 | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 5 | 4 | 1
insomnia (Psychiatric disorders) | 1 | 3 | 1
Depression (Psychiatric disorders) | 0 | 0 | 2
Depressed Mood (Psychiatric disorders) | 0 | 2 | 0
Major Depression (Psychiatric disorders) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 5 | 3 | 3
Dizziness (Nervous system disorders) | 1 | 2 | 1
Palpations (Cardiac disorders) | 0 | 0 | 2
oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 5
Erythema (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
fatigue (General disorders) | 1 | 1 | 2
Odema Peripheral (General disorders) | 1 | 0 | 2
Odema (General disorders) | 0 | 0 | 2
Blood Pressure Increased (Investigations) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other